CLINICAL TRIAL: NCT04093999
Title: Nerve Coaptation Improves the Sensory Recovery of the Breast in DIEP Flap Breast Reconstruction
Brief Title: Sensory Nerve Coaptation in DIEP Flap Breast Reconstruction
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Rene van der Hulst, Head of the Plastic Surgery department, Maastricht University Medical Center
Other Study IDs: METC 16 - 4 - 147
Record Dates: First submitted 2019-09-17; First posted 2019-09-18 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: Breast reconstruction; DIEP flap; Sensory recovery; Breast sensation; Nerve coaptation
MeSH Terms: conditions — Breast Neoplasms | interventions — Nerve Transfer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Innervated DIEP flaps: Patients in this group underwent immediate or delayed, unilateral or bilateral DIEP flap breast reconstruction with additional sensory nerve coaptation.
  Interventions: Procedure: Sensory nerve coaptation
- Noninnervated DIEP flaps: Patients in this group underwent immediate or delayed, unilateral or bilateral DIEP flap breast reconstruction without sensory nerve coaptation.

INTERVENTIONS:
Procedure: Sensory nerve coaptation — A recipient sensory nerve branch of the 11th-12th intercostal nerve was reattached to a donor nerve in the chest area. The anterior cutaneous branch of the second or third intercostal nerve was used as the donor nerve. Direct, end-to-end nerve coaptation was performed.
  Other Names: Neurotization; Reinnervation; Neurorrhaphy
  Groups: Innervated DIEP flaps

SUMMARY:
Restoring the sensation of the breast becomes increasingly recognized as a critical part of autologous breast reconstruction. A prospective study was conducted of all patients who underwent either innervated or non-innervated deep inferior epigastric perforator (DIEP) flap breast reconstruction in Maastricht University Medical Center between August 2016 and August 2018 and who returned between for a follow-up visit between the start of the study and August 2019. Semmes-Weinstein monofilaments were used for sensory testing of the breast.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years or older
* Unilateral or bilateral DIEP flap breast reconstruction
* Returned for follow-up between August 2016 and August 2019
* Informed consent

Exclusion Criteria:

* Total flap loss complication
* Flaps that required a take-back
* Follow-up less than six months postoperatively
* Only one postoperative measurement at less than 12 months follow-up
* Mixed reconstructions: an innervated breast reconstruction on one side and a noninnervated breast reconstruction on the other side

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients of 18 years or older.
Study Population: In this prospective study, patients who underwent an innervated or noninnervated DIEP flap breast reconstruction between August 2016 and August 2018 at Maastricht University Medical Center in the Netherlands were included if they returned for follow-up between August 2016 and August 2019.
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Mean monofilament value as a measure for the sensory recovery of the reconstructed breast | Through study completion up to 36 months postoperatively
  The sensory recovery of the breast to touch was tested at different follow-up moments after the initial surgery. Semmes-Weinstein monofilaments were used for sensory testing. Nine areas of the breast, indicating native skin and flap skin, were tested. Mean monofilament values were calculated for each area and compared between groups.

SECONDARY OUTCOMES:
Mean monofilament value as a measure for the sensory recovery of the reconstructed breast | Through study completion up to 36 months postoperatively
  The sensory recovery of the donor site to touch was tested at different follow-up moments after the initial surgery. Semmes-Weinstein monofilaments were used for sensory testing. Four areas of the donor site were tested, two areas above and two areas below the scar. Mean monofilament values were calculated for the total donor site and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: René van der Hulst, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No